CLINICAL TRIAL: NCT00112125
Title: Evaluation of the Safety and Efficacy of the OPTIMIZER System With Active Fixation Leads in Subjects With Heart Failure Resulting From Systolic Dysfunction: FIX-HF-5
Brief Title: Evaluation of the Safety and Effectiveness of the OPTIMIZER System in Subjects With Heart Failure: FIX-HF-5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #IDPT 2003-07-C; FIX-HF-5 (Other: Impulse Dynamics)
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure, Congestive
Keywords: cardiac contractility modulation; heart failure; cardiopulmonary exercise test; chronic heart disease
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimizer System + Optimal medical treatment (Experimental): Optimizer System implanted and cardiac contractility modulation therapy activated.
  Interventions: Device: OPTIMIZER System
- Optimal medical treatment (No Intervention): Treatment with optimal medical therapy only.

INTERVENTIONS:
Device: OPTIMIZER System
  Arms: Optimizer System + Optimal medical treatment

SUMMARY:
The purpose of this study is to determine whether treatment with the OPTIMIZER System is safe and effective in patients with moderate to severe heart failure symptoms.

DETAILED DESCRIPTION:
IMPULSE Dynamics' FIX HF 5 US Study is a prospective, multi-center, study to evaluate the safety and efficacy of cardiac contractility modulation (CCM) signals delivered by the implantable OPTIMIZER™ System in patients with NYHA class III/IV heart failure. The study will involve the recruitment of approximately 420 subjects at a total of up to 50 sites nationwide.

Those subjects who fulfill all inclusion and exclusion criteria based upon baseline test results will be randomized to receive the OPTIMIZER™ System or to a control group. All subjects randomized will be followed for 1 year and shall receive the same study related assessments throughout the course of the study. In addition, all subjects will continue to receive optimal medical therapy for the treatment of their heart failure.

The primary efficacy assessment consists of a change in exercise tolerance measured by cardiopulmonary exercise testing at baseline and 6 months. Safety variables, such as the rate and cause of hospitalizations or death, shall be collected in both groups and shall be compared at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 years of age or older
* Subjects who are either male or female
* Subjects who have a baseline ejection fraction of 35% or less by echocardiography.
* Subjects who have been treated for heart failure for at least 90 days (including treatment with a β-blocker for at least 90 days unless the patient is intolerant) and are in New York Heart Association functional Class III or IV at the time of enrollment.
* Subjects receiving appropriate, stable medical therapy during the 30 days prior to enrollment for treatment of heart failure, consisting of the appropriate doses of diuretics, ACE-inhibitor or angiotensin II receptor blocker and β-blocker. Stable is defined as no more than a 100% increase or 50% decrease in dose.
* Subjects who, in the opinion of the Principle Investigator (based on the current guidelines for clinical practice), have a clinical indication for an implanted cardiac defibrillator (ICD) and/or pacemaker, must have an existing device or agree to undergo implantation of such a device unless the patient refuses to undergo the implantation of such device for personal reasons.
* Subjects who are willing and able to return for all follow-up visits.

Exclusion Criteria:

* Subjects whose baseline VO2,max is <9 ml 02/min/kg.
* Subjects who have a potentially correctible cause of heart failure, such as valvular heart disease or congenital heart disease.
* Subjects who have clinically significant angina pectoris, consisting of angina during daily life (i.e., Canadian Cardiovascular Society Angina score of II or more), an episode of unstable angina within 30 days of enrollment, or angina and/or electrocardiography (ECG) changes during exercise testing performed during baseline evaluation.
* Subjects who have been hospitalized for heart failure which required the use of inotropic support within 30 days of enrollment.
* Subjects who have a clinically significant amount of ambient ectopy, defined as more than 8,900 premature ventricular complexes (PVCs) per 24 hours on baseline Holter monitoring.
* Subjects who have chronic atrial fibrillation or chronic atrial flutter or those cardioverted within 30 days of enrollment.
* Subjects whose exercise tolerance is limited by a condition other than heart failure (e.g., angina, chronic obstructive pulmonary disease [COPD], peripheral vascular disease, orthopedic or rheumatologic conditions) or who are unable to participate in a 6-minute walk or a cardiopulmonary stress test.
* Subjects who are scheduled for a coronary artery bypass graft (CABG) or a percutaneous transluminal coronary angioplasty (PTCA) procedure, or who have undergone a CABG procedure within 90 days or a PTCA procedure within 30 days of enrollment.
* Subjects who have a biventricular pacing system or who have an accepted indication for such a device.
* Subjects who have had a myocardial infarction within 90 days of enrollment.
* Subjects who have mechanical tricuspid or aortic valves.
* Subjects who have a prior heart transplant.
* Subjects who are participating in another experimental protocol.
* Subjects who are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2005-02 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Burkhoff, M.D, Ph.D., Study Director — Impulse Dynamics
Locations (1):
- Impulse Dynamics, Orangeburg, New York, United States

REFERENCES:
- [Background] Burkhoff D, Shemer I, Felzen B, Shimizu J, Mika Y, Dickstein M, Prutchi D, Darvish N, Ben-Haim SA. Electric currents applied during the refractory period can modulate cardiac contractility in vitro and in vivo. Heart Fail Rev. 2001 Jan;6(1):27-34. doi: 10.1023/a:1009851107189. No abstract available. PMID 11248765
- [Background] Ellison K. Nonexcitatory stimulation: 2002: a pace odyssey. J Cardiovasc Electrophysiol. 2002 Jul;13(7):696-7. doi: 10.1046/j.1540-8167.2002.00696.x. No abstract available. PMID 12139295
- [Background] Marrouche NF, Pavia SV, Zhuang S, Kim YJ, Tabata T, Wallick D, Saad E, Abdul-Karim A, Schweikert R, Saliba W, Tchou P, Natale A. Nonexcitatory stimulus delivery improves left ventricular function in hearts with left bundle branch block. J Cardiovasc Electrophysiol. 2002 Jul;13(7):691-5. doi: 10.1046/j.1540-8167.2002.00691.x. PMID 12139294
- [Background] Mohri S, He KL, Dickstein M, Mika Y, Shimizu J, Shemer I, Yi GH, Wang J, Ben-Haim S, Burkhoff D. Cardiac contractility modulation by electric currents applied during the refractory period. Am J Physiol Heart Circ Physiol. 2002 May;282(5):H1642-7. doi: 10.1152/ajpheart.00959.2001. PMID 11959626
- [Background] Morita H, Suzuki G, Haddad W, Mika Y, Tanhehco EJ, Sharov VG, Goldstein S, Ben-Haim S, Sabbah HN. Cardiac contractility modulation with nonexcitatory electric signals improves left ventricular function in dogs with chronic heart failure. J Card Fail. 2003 Feb;9(1):69-75. doi: 10.1054/jcaf.2003.8. PMID 12612875
- [Background] Mohri S, Shimizu J, Mika Y, Shemer I, Wang J, Ben-Haim S, Burkhoff D. Electric currents applied during refractory period enhance contractility and systolic calcium in the ferret heart. Am J Physiol Heart Circ Physiol. 2003 Apr;284(4):H1119-23. doi: 10.1152/ajpheart.00378.2002. Epub 2002 Nov 21. PMID 12446280
- [Background] Sabbah HN, Haddad W, Mika Y, Nass O, Aviv R, Sharov VG, Maltsev V, Felzen B, Undrovinas AI, Goldstein S, Darvish N, Ben-Haim SA. Cardiac contractility modulation with the impulse dynamics signal: studies in dogs with chronic heart failure. Heart Fail Rev. 2001 Jan;6(1):45-53. doi: 10.1023/a:1009855208097. PMID 11248767
- [Background] Pappone C, Rosanio S, Burkhoff D, Mika Y, Vicedomini G, Augello G, Shemer I, Prutchi D, Haddad W, Aviv R, Snir Y, Kronzon I, Alfieri O, Ben-Haim SA. Cardiac contractility modulation by electric currents applied during the refractory period in patients with heart failure secondary to ischemic or idiopathic dilated cardiomyopathy. Am J Cardiol. 2002 Dec 15;90(12):1307-13. doi: 10.1016/s0002-9149(02)02868-0. PMID 12480039
- [Derived] Abraham WT, Burkhoff D, Nademanee K, Carson P, Bourge R, Ellenbogen KA, Parides M, Kadish A; FIX-HF-5 Investigators and Coordinators. A randomized controlled trial to evaluate the safety and efficacy of cardiac contractility modulation in patients with systolic heart failure: rationale, design, and baseline patient characteristics. Am Heart J. 2008 Oct;156(4):641-648.e1. doi: 10.1016/j.ahj.2008.05.019. PMID 18926146

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group (OMT): Optimal medical treatment (OMT). Subjects receiving appropriate, stable medical therapy during the 30 days prior to enrollment for treatment of heart failure, consisting of the appropriate doses of diuretics, ACE-inhibitor or angiotensin II receptor blocker and B-blocker.
- Treatment (CCM + OMT): Treatment group: Subjects receiving OMT and cardiac contractility modulation therapy with the Optimizer System.
Period: Overall Study
Arm/Group | Control Group (OMT) | Treatment (CCM + OMT)
Started | 213 | 215
Completed | 189 | 193
Not Completed | 24 | 22

BASELINE CHARACTERISTICS:
Groups:
- Treatment (OMT + CCM): Treatment group: Subjects receiving OMT and cardiac contractility modulation therapy with the Optimizer System.
- Total: Total of all reporting groups
Arm/Group | Control Group (OMT) | Treatment (OMT + CCM) | Total
Number analyzed (Participants) | 213 | 215 | 428
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (12.2) | 58.1 (12.8) | 58.35 (12.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 57 | 119
  Male | 151 | 158 | 309
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 36 | 81
  White | 142 | 154 | 296
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 18 | 39
Region of Enrollment [Number; unit: participants]
  United States | 213 | 215 | 428
Peak VO2 [Mean (Standard Deviation); unit: ml/kg/min] | 14.71 (2.92) | 14.74 (3.06) | 14.725 (2.99)
6 Minute Hall Walk Distance [Mean (Standard Deviation); unit: meters] | 324 (92.4) | 326.4 (82.1) | 325.2 (7.28)
NYHA Class III [Count of Participants; unit: Participants] — Class I: Ordinary physical activity does not cause undue dyspnea or fatigue.
  Class II: Comfortable at rest. Ordinary physical activity results in dyspnea or fatigue.
  Class III: Comfortable at rest. Less than ordinary physical activity results in dyspnea or fatigue.
  Class IV: Symptoms of heart failure may be present even at rest. If any physical activity is undertaken, discomfort is increased.
  Participants | 183 | 196 | 379
NYHA Class IV [Count of Participants; unit: Participants] — Class I: Ordinary physical activity does not cause undue dyspnea or fatigue.
  Class II: Comfortable at rest. Ordinary physical activity results in dyspnea or fatigue.
  Class III: Comfortable at rest. Less than ordinary physical activity results in dyspnea or fatigue.
  Class IV: Symptoms of heart failure may be present even at rest. If any physical activity is undertaken, discomfort is increased.
  Participants | 29 | 19 | 48
MLWHFQ score [Mean (Standard Deviation); unit: Score on a scale] — Minnessotta Living with Heart Failure Questionnaire score. There are 21 questions completed by the participant, with each response on a scale of 0-5. The total score ranges from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life.
  Score on a scale | 57.4 (22.6) | 60.5 (23) | 58.95 (0.282)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Endpoint: Ventilatory Anerobic Threshold (VAT)
Description: Number of participants with improvement in exercise tolerance at 24 weeks compared to baseline, as quantified by VO2 at ventilatory anerobic threshold (VAT) measured on cardiopulmonary exercise stress testing (CPX), and evaluated by a blinded core lab.
  Note: An individual subject is considered a responder if VAT increases by ≥20% at 24 weeks compared to their respective baseline value.
Time Frame: 24 weeks
Population: Intention to treat (ITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (OMT) | Treatment (CCM + OMT)
Number analyzed (Participants) | 213 | 215
Participants | 28 | 38
Statistical Analysis 1: Comparison: Control Group (OMT) vs Treatment (CCM + OMT); Test type: Non-Inferiority — The primary safety analysis was a test of the non-inferiority of CCM therapy compared to OMT with respect to the proportion of subjects experiencing death or hospitalization within 50 weeks using the Blackwelder non-inferiority test12 with a prespecified non-inferiority margin of 0.125; p = 0.31, Fisher Exact

2. Primary Outcome: Safety Endpoint: Composite All-cause Mortality and All-cause Hospitalizations
Description: The proportion of patients experiencing a composite event of all-cause mortality and all-cause hospitalizations evaluated at 50-weeks
Time Frame: 50-weeks
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (OMT) | Treatment (CCM + OMT)
Number analyzed (Participants) | 213 | 215
Participants | 103 | 112
Statistical Analysis 1: Comparison: Control Group (OMT) vs Treatment (CCM + OMT); Test type: Non-Inferiority — The noninferiority margin was selected to be 12.5% and α was set at .05, which resulted in a sample size of 198 subjects per group. A percentage of subjects (∼7%) were expected to be lost to followup, so that a total sample size of 428 subjects (214 per group) was selected; p = 0.125, Blackwelder

3. Secondary Outcome: Peak VO2
Description: Number of participants with improvement in peak VO2 measured on cardiopulmonary exercise stress testing (CPX), and evaluated by a blinded core lab.
  Note: An individual subject is considered a responder if peak VO2 increases by ≥20% at 24 weeks compared to their respective baseline value.
Time Frame: 24 weeks
Population: Completed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (OMT) | Treatment (CCM + OMT)
Number analyzed (Participants) | 168 | 179
Participants | 23 | 31

4. Secondary Outcome: New York Heart Association (NYHA) Functional Classification
Description: Number of participants with improvement in heart failure symptoms as quantified by a blinded clinician using the New York Heart Association (NYHA) functional classification at 24 weeks compared to baseline. The NYHA Class ranges from I - IV, with a lower class indicating a better status.
  Note: An individual subject is considered a responder if the NYHA class decreases by ≥ 1 at 24 weeks compared to their respective baseline class.
Time Frame: 24 weeks
Population: Completed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (OMT) | Treatment (CCM + OMT)
Number analyzed (Participants) | 183 | 191
Participants | 63 | 94

5. Secondary Outcome: Minnesota Living With Heart Failure (MLWHF) Questionnaire
Description: Number of subjects will improvement in quality of life at 24 weeks compared to baseline, as assessed by the Minnesota Living with Heart Failure (MLWHF) Questionnaire. The MLWHFQ score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life.
  Note: An individual subject is considered a responder if the MLWHFQ score decreases by ≥10 points at 24 weeks compared to their respective baseline score.
Time Frame: 24 weeks
Population: Completed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (OMT) | Treatment (CCM + OMT)
Number analyzed (Participants) | 184 | 196
Participants | 77 | 110

6. Secondary Outcome: Six Minute Hall Walk (6MW) Test
Description: Number of subjects with improvement in exercise tolerance at 24 weeks compared to baseline, as assessed by the the six minute hall walk (6MW) test.
  Note: An individual subject is considered a responder with >40-meter increase in distance walked at 24 weeks compared to their respective baseline distance.
Time Frame: 24 weeks
Population: Completed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (OMT) | Treatment (CCM + OMT)
Number analyzed (Participants) | 173 | 190
Participants | 51 | 65

ADVERSE EVENTS:
Time Frame: 50-weeks
Arm/Group | Control Group (OMT) | Treatment (CCM + OMT)
All-Cause Mortality (participants affected / at risk) | 7/212 | 13/210
Serious Adverse Events (participants affected / at risk) | 115/212 | 129/210
Other Adverse Events (participants affected / at risk) | 135/212 | 152/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (OMT) (N=212) | Treatment (CCM + OMT) (N=210)
General Cardiopulmonary Event (Cardiac disorders) | 46 (58) | 42 (60)
Arrhythmia (Cardiac disorders) | 25 (30) | 29 (40)
General Medical (General disorders) | 54 (81) | 63 (98)
ICD or Pacemaker System Malfunction (Cardiac disorders) | 6 (7) | 11 (13)
Localized Infection (Infections and infestations) | 29 (36) | 27 (33)
Worsening Heart Failure (Cardiac disorders) | 50 (85) | 50 (72)
Bleeding (Blood and lymphatic system disorders) | 8 (8) | 6 (8)
Sepsis (Infections and infestations) | 2 (2) | 10 (11)
Neurologic Dysfunction (Nervous system disorders) | 12 (14) | 3 (3)
Thromboembolism (Vascular disorders) | 5 (5) | 3 (3)
OPTIMIZER lead fracture (Surgical and medical procedures) | 0 (0) | 3 (3)
OPTIMIZER RV lead dislodgement (Surgical and medical procedures) | 0 (0) | 6 (6)
IPG problem/change (Surgical and medical procedures) | 0 (0) | 1 (2)
OPTIMIZER RA lead dislodgement (Surgical and medical procedures) | 0 (0) | 5 (6)
OPTIMIZER pocket dehiscence/erosion (Surgical and medical procedures) | 0 (0) | 3 (3)
OPTIMIZER pocket infection (Infections and infestations) | 0 (0) | 2 (2)
OPTIMIZER pocket stimulation (Surgical and medical procedures) | 0 (0) | 2 (2)
Lead perforation (Surgical and medical procedures) | 0 (0) | 2 (2)
OPTIMIZER pocket bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sensation due to CCM (Surgical and medical procedures) | 0 (0) | 2 (2)
Extracardiac stimulation (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (OMT) (N=212) | Treatment (CCM + OMT) (N=210)
General Cardiopulmonary Event (Cardiac disorders) | 19 (21) | 41 (55)
Arrhythmias (Cardiac disorders) | 13 (16) | 26 (29)
Worsening Heart Failure (Cardiac disorders) | 29 (35) | 32 (35)
Localized Infection (Infections and infestations) | 41 (50) | 51 (63)
General Medical (General disorders) | 86 (167) | 105 (193)

LIMITATIONS AND CAVEATS:
The primary endpoint was not validated for use in HF trials (VAT, responder analysis, responder = 20% increase). VAT was missing or indeterminant in 30% of subjects despite use of 2 blinded core labs. ITT analysis required 10 levels of imputation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-08-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT00112125/Prot_SAP_ICF_000.pdf